CLINICAL TRIAL: NCT05950594
Title: Prospective Study of Image and Blood-derived Biomarkers to Predict Metastasis in Soft-tissue Sarcomas
Brief Title: IVIM & OLINK in Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-5436
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy — Standard of care pre-operative radiotherapy
Other: Surgery — Standard of care definitive surgery

SUMMARY:
The hypoxia > metastasis axis suggests that a DWI-based biomarker of hypoxia incorporating IVIM may be able to predict metastasis in STS patients, ultimately enabling stratification for personalized treatments at the time of diagnostic (MR) imaging, without adding an excessive burden to the patient or clinical workflow (typical DWI/IVIM sequences can be acquired acquired in approximately 5 minutes).

DETAILED DESCRIPTION:
Tumour hypoxia has been implicated as a major driver in STS metastatic dissemination. Despite this, patients are not routinely assessed for hypoxia, largely due to the cost and difficulty involved. PET hypoxia imaging using Fluorine-18-labelled nitroimidazole-based agents such as fluoroazomycin arabinoside (FAZA) provide non-invasive in vivo quantification of hypoxia [5], including in STS. The expense and unproven clinical value of these agents and the long times between their injection and PET scanning (typically, two hours) has limited the uptake of PET-hypoxia imaging as a routine screening modality. In contrast, magnetic resonance imaging (MRI) is standard for diagnosis of STS and is a routine part of the radiation therapy workflow due to its superior contrast between tumour and surrounding normal tissue. In addition, diffusion-weighted magnetic resonance imaging (DWI) can quantify physiological tumour properties such as cellularity and perfusion that may provide information about tumour biology, including hypoxia.

Hypoxia results from the interplay between oxygen demand (oxygen consumption rate) and supply (perfusion). Hypothesizing that oxygen consumption increases with increasing cellularity, Hompland and colleagues demonstrated that a biomarker derived from IVIM measurements could predict hypoxia in prostate, breast, and cervical cancer patients. An ongoing prospective imaging study of hypoxia in STS patients at Princess Margaret is investigating the capacity of FAZA to image hypoxia in STS and develop correlative DWI (IVIM)-based biomarkers of hypoxia on a combined PET/MRI scanner.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ability to understand and the willingness to sign a written informed consent document
* Grade 2 or 3 soft tissue sarcoma greater than 5 cm in largest dimension

Exclusion Criteria:

* Contraindication to MRI scan as per current institutional guidelines (for patients requiring MRI)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Identify image-derived, plasma-derived biomarkers of hypoxia | 3 years
  Image-derived, plasma-derived biomarkers of hypoxia (such as HIF-1alpha, VEGF, osteopontin) acquired before radiation therapy will be assessed for correlation to distant metastasis-free survival.

SECONDARY OUTCOMES:
Hypoxia in plasma | 3 years
  Correlation between the relative concentration of circulating protein biomarkers of hypoxia detected in plasma using proximity-extension assays to hypoxic fraction as calculated by MR imaging and to distant metastasis-free survival.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada